CLINICAL TRIAL: NCT01674387
Title: Lu's Acupuncture Protocol for Chronic Neck Pain
Brief Title: Clinical Study on Electroacupuncture Therapy for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Principal Investigator, Jian Pei,MD, MD,professor, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 64385700; ZYSNXD-CCHPGC-JD-007 (Other: Shanghai Municipal Commission of Health and Family Planning)
Record Dates: First submitted 2012-08-16; First posted 2012-08-28 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Neck Pains
Keywords: electroacupuncture therapy; neck pain; McGill Pain Questionnaire; Acupuncture Therapy; Electroacupuncture; Meridians
MeSH Terms: conditions — Neck Pain | interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture (Experimental): 56 patients (the EA group) receive the acupuncture treatment at nine acupuncture points: Dazhui (GV14), bilateral Jianzhongshu (SI15), bilateral Jingbailao (EX HN15), bilateral cervical Jiaji (EX-B2),and two trigger points.Bilateral Jianzhongshu (SI15) and Jiaji (EX-B2) receive the electro acupuncture treatment, with dilatational wave. All the needles retained for 20 minutes, one treatment every other day, 10 times a course, and the treatment assessed after a course.
  Interventions: Device: acupuncture
- comprehensive treatment (Other): Other 56 patients (the matched group) receive the comprehensive treatment, including traction and TENS(Transcutaneous Electrical Nerve Stimulation) therapy. Each treatment 20 minutes, one treatment every other day, 10 times a course, and the treatment assessed after a course.
  Interventions: Other: comprehensive treatment

INTERVENTIONS:
Device: acupuncture — 56 patients (the EA group) receive the acupuncture treatment at nine acupuncture points: Dazhui (GV14), bilateral Jianzhongshu (SI15), bilateral Jingbailao (EX HN15), bilateral Jiaji (EX-B2) of cervical positive reaction plane (taking two pairs). Besides, bilateral Jianzhongshu (SI15) and bilateral Jiaji (EX-B2) receive the electro acupuncture treatment, with dilatational wave. All the needles retained for 20 minutes, one treatment every other day, 10 times a course, and the treatment assessed after a course.
  Other Names: electroacupuncture
  Arms: acupuncture
Other: comprehensive treatment — Other 56 patients (the matched group) receive the comprehensive treatment, including traction and TENS therapy. Each treatment 20 minutes, one treatment every other day, 10 times a course, and the treatment assessed after a course.
  Arms: comprehensive treatment

SUMMARY:
Purpose of this test is to observe and objectively evaluate electroacupuncture (EA) therapy on the clinical efficacy in patients with chronic neck pain, and provide a reliable clinical basis for the chronic neck pain treatment and evaluation of efficacy.

DETAILED DESCRIPTION:
According to statistics, the incidence of chronic neck pain has significantly increased year by year, particularly tending to younger people, as social competition increase fiercely and the pace of people's daily work and life accelerate. Studying the effective treatment and prevention of chronic neck pain has obvious medical, social and economic significance. Purpose of this trial is to observe and objectively evaluate electroacupuncture (EA) therapy on the clinical efficacy in patients with chronic neck pain, and provide a reliable clinical basis for the chronic neck pain treatment and evaluation of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age of a subject is older than 18 and is younger than 65.
2. With more than 3 months history of neck pain.
3. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. With serious protopathy or disease ofcardiovascular,liver,renal,gastrointestinal, hematological systems and so on.
2. Psychotic，patients with allergic constitution or easily getting infected or bleeding.
3. Patients have used drugs for preventing neck pain in the last four weeks.
4. Pregnant women or women in lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
chronic neck pain-the Neck Pain Scale (NPQ) | 20 days(One course)
the short-form McGill Pain Questionnaire | 20 days(One course)
the SF-36 Health Questionnaire combined with Neck Disability Index (NDI). | 20 days(one course)

SECONDARY OUTCOMES:
chronic neck pain-the Neck Pain Scale (NPQ) | one month after a course.
the short-form McGill Pain Questionnaire | one month after a course
the SF-36 Health Questionnaire combined with Neck Disability Index (NDI). | one months after a course

CONTACTS AND LOCATIONS:
Overall Officials: Jian Pei, MD, Study Director — Longhua Hospital; Qinhui Fu, MD, Principal Investigator — Longhua Hospital; Jia Yan, MM, Principal Investigator — Shanghai Univercity of TCM